CLINICAL TRIAL: NCT00293514
Title: An Open, Randomised, Prospective, Multi-centre, Parallel-group Trial of TachoSil Versus Standard Surgical Treatment in Patients Undergoing Pulmonary Lobectomy for Lung Malignancy and Requiring Treatment for Air Leakage
Brief Title: TachoSil Versus Standard Surgical Treatment for Air Leakage in Pulmonary Lobectomy (TC-021-IM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-021-IM; 2004-002380-24
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-02

CONDITIONS: Pulmonary Diseases; Intraoperative Complications
Keywords: standard surgical treatment for air leakage in pulmonary lobectomy
MeSH Terms: conditions — Lung Diseases; Intraoperative Complications | interventions — Fibrinogen; Thrombin; TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fibrinogen (human) + thrombin (human) (TachoSil)

SUMMARY:
The purpose of this study is to compare the sealing efficacy and safety of TachoSil® (hereafter referred to as TachoSil) versus standard surgical treatment as the secondary management of intra-operative pulmonary air leakage after a lobectomy in subjects with lung malignancies with or without metastases.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of lung malignancy with or without metastases may be included in the trial if the entry criteria apply.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Duration of post-operative air leakage: assessment on the evening of the day of operation (Day 0) and then subsequently twice daily (on morning and evening shifts)

SECONDARY OUTCOMES:
Reduction of intra-operative air leakage intensity after first application of trial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (1):
- Nycomed, Roskilde, Denmark